CLINICAL TRIAL: NCT02906631
Title: Epidemiology and Prognosis of Encephalitis in Intensive Care
Acronym: ENCEPHALITICA
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: AOR 15096
Record Dates: First submitted 2016-09-01; First posted 2016-09-20 (Estimated); Last update posted 2024-03-20 (Actual); Status verified 2024-03

CONDITIONS: Encephalitis
Keywords: encephalitis,; neurologic outcomes of all-cause encephalitis in intensive care unit; outcome, intensive care unit
MeSH Terms: conditions — Encephalitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood and cerebrospinal fluid samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients admitted to the ICU for AE: Adult patients with all-cause encephalitis admitted to an intensive care unit.

SUMMARY:
Introduction: Acute encephalitis (AE) is a severe neurological disorder associated with significant morbidity and mortality. Approximately 50% of patients with AE require ICU admission because of coma, seizures or acute respiratory failure. Determinants of neurological prognosis in these patients are not known.

Objectives:

Main objective: To identify determinants of outcome in adult patients admitted to the ICU; Secondary objectives: a) To study the impact of diagnostic studies (Brain MRI, CSF analysis, EEG) on neurologic outcome; b) to describe the epidemiology of patients admitted to the ICU with AE; c) to study the impact of early appropriate therapy on neurologic outcomes; d) to describe morbidity and mortality associated with AE at 90 days and 1 year following diagnosis.

Methods: prospective observational multicenter study in French ICUs. All patients admitted to the ICU for probable or confirmed AE (2013 IDSA criteria)with a Glasgow coma scale score < or =to 13 will be eligible for inclusion. Factors associated with a poor prognosis at 90 days will be identified by multivariable logistic regression analysis.

Duration of study: 30 months (recruitment 18 months, follow-up 12 months).

Patients: 300 patients

Endpoints:

* Primary endpoint: The primary endpoint is the modified Rankin scale score 90 days following onset of abnormal status (GCS < or =13). This score will be determined by contacting the patient. A poor outcome will be defined as a mRS >2 at 90 days.
* Secondary endpoints: a) neurological findings within 7 days following onset of altered mental status; b) abnormal findings on diagnostic studies (MRI, EEG, CSF analysis) within7 days following onset of altered mental status; c) Time between onset of altered mental status and completion of diagnostic studies; d)Time between onset of altered mental status and start of appropriate specific therapy; e) neurologic outcomes at 1 year mRS score and extended Glasgow outcome scale (GOS); f) causes of death in non-survivors at 1 year; g) quality of life and posttraumatic stress at 1 year: IADL and SF36 scales;

DETAILED DESCRIPTION:
Acute encephalitis (AE) is a serious condition associated with significant morbidity and mortality. Patients require ICU admission in 60 % of cases, mainly because of neurological symptoms (coma, seizures) or acute respiratory failure.

The etiological profile of AE has changed considerably in recent years, with the emergence of new pathogens and the description of new immune-mediated causes (acute disseminated encephalomyelitis (ADEM), autoimmune limbic encephalitis) that require urgent specific therapies. Furthermore, despite extensive investigations, the proportion of cases of unknown cause remains high.

In-ICU care of patients with AE is a difficult task, given the diversity of etiologies and clinical presentations. Furthermore, additional studies such as magnetic resonance imaging (MRI) can be challenging to obtain in this population. Finally, there are no specific recommendations on the management and prognostic assessment of patients admitted to the ICU with AE.

Present available data on the prognosis of patients with AE include both adult and pediatric cases, and focuses only on AE with identified causes. Prognosis of encephalitis in adult patients requiring ICU admission has been previously described only in retrospective single centre cohorts. To date, no prospective multicenter study on AE has been conducted in the specific population of adult critically ill patients. Furthermore, data on the diagnostic and prognostic contributions of magnetic resonance imaging (MRI) and electroencephalography studies in these patients are lacking The development of guidelines for standardized care in critically ill AE patients is needed, and will include management of early life support, prompt and exhaustive etiologic investigations, early administration of specific treatments and assessment of neurological prognosis. This study, which will focus on prognostic evaluation of severe AE in adults, appears crucial to support the development of such guidelines.

Patients admitted to ICU for a suspicion of AE (acute encephalopathy and CSF pleocytosis > 5 cells / microliter) will be eligible for inclusion.

Patients admitted to ICU for a suspicion of AE (acute encephalopathy and CSF pleocytosis > 5 cells / microliter) will be eligible for inclusion. Eligible patients will be included if they fulfil the IDSA 2013 diagnostic criteria for ""probable"" or ""confirmed"" encephalitis (see inclusion criteria). In patients without an obvious etiological diagnosis, an algorithm will be suggested to investigators to guide etiological investigations, according to the most recent recommendations (IDSA 2013). Aetiology of encephalitis will be described according to a priori-defined categories: 1) viral causes, 2) immune-mediated-causes, 3) bacterial or fungal meningitis with secondary encephalitic features, 4) undetermined causes. For each included patient, CSF and plasma samples will be stored at -80°C. A biobank will be created for subsequent analyses (etiological diagnosis, prognostic biomarkers). Outcomes will be assessed at 90 days and 365 days by contacting the patient or his relatives. The primary outcome is the score on the modified Rankin scale, which will be assessed 90 days after inclusion. Independent predictors of functional outcomes will be determined by multivariate logistic regression analysis.

ELIGIBILITY:
Inclusion criteria:

* Altered mental status, delirium, or personality changes for a duration > or = 24 h
* At least 2 of the following: 1) fever (>38°C) within 72 hours before or following hospital admission; 2) new-onset seizures; 3) new-onset focal signs; 4) CSF pleocytosis > 5 cell / microl; 5) brain parenchyma abnormalities on neuroimaging compatible with the diagnosis of encephalitis; 6) EEG abnormalities compatible with the diagnosis of encephalitis.
* Altered mental status with a GCS < or =13 without sedation, or GCS < or =13 before sedation administration in sedated patients
* CSF analysis performed
* Brain imaging performed (CT/MRI)
* Age >18

Exclusion criteria:

* Time between the first hospitalization for neurologic symptoms in relation with encephalitis and ICU admission > 21 days
* Purulent bacterial meningitis diagnosed by direct examination or CSF analysis
* Isolated brain abscess.
* Febrile encephalopathy associated with another diagnosis
* Predicted time in ICU < or = 24 hours
* Opposition of close-of-kin, if present at the inclusion, for patient participation in research.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to ICU for a suspicion of AE (acute encephalopathy and CSF pleocytosis > 5 cells / microliter) will be eligible for inclusion.
Sampling Method: Non-Probability Sample
Enrollment: 350 (Actual)
Dates: Start 2017-10-27 (Actual); Primary Completion 2023-04-20 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
Neurological status on the modified Rankin scale | 90 days
  The primary outcome measure is the modified Rankin scale score 90 days following onset of abnormal status (defined by a GCS score< or =13). This score will be determined by contacting the patient or his relatives. A poor outcome will be defined as a mRS >2 at 90 days.

SECONDARY OUTCOMES:
Biological data within 7 days following onset of altered mental status | 7 days
State of consciousness defined by the Glasgow Coma Scale within 7 days following onset of altered mental status | 7 days
Patient's comorbidity measured by Charlson Comorbidity Index | 7 days
Presence of focal neurological deficit within 7 days following onset of altered mental status | 7 days
Presence of thermal dysregulation within 7 days following onset of altered mental status | 7 days
Presence of seizures within 7 days following onset of altered mental status | 7 days
Magnetic resonance imaging anomalies within 7 days following onset of altered mental status | 7 days
Electrophysiologic anomalies within 7 days following onset of altered mental status | 7 days
Time between onset of altered mental status and cerebrospinal fluid analysis | one year
Time between onset of altered mental status and brain magnetic resonance imaging study | one year
Time between onset of altered mental status and electroencephalogram study | one year
Time between onset of altered mental status and completion of diagnostic studies (CSF analysis, MRI, EEG) | one year
Number of patients with primitive acute encephalitis (AE) | 7 days
  Number of patients with infectious causes leading to primitive AE
Number of patients with infectious causes leading to meningitis with secondary encephalitic features | 7 days
Number of patients with immune-mediated causes of encephalitis | 7 days
Number of patients with other infectious causes of encephalitis | 7 days
Proportion of patients with appropriate specific therapy | 7 days
Time between onset of altered mental status and appropriate specific therapy | one year
Neurological status on the modified Rankin scale | 365 days
  This score will be determined by contacting the patient or his relatives.
Hospital anxiety and depression scale (HAD) | 365 days
Quality of life measured by SF36 scale | 365 days
INSTRUMENTAL ACTIVITIES OF DAILY LIVING SCALE (IADL) | 365 days
Neurological prognosis on the extended Glasgow outcome scale | 365 days

CONTACTS AND LOCATIONS:
Overall Officials: Romain Sonneville, M.D. Ph.D., Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital Bichat-Claude Bernard, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided